CLINICAL TRIAL: NCT04311970
Title: Pilot Study of EsoCheck Compared to Biopsies and Brush Cytology During Endoscopy for Evaluation of Eosinophilic Esophagitis.
Brief Title: Pilot Study of Esocheck in Eosinophilic Esophagitis
Acronym: EoE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Lucid Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 833846
Record Dates: First submitted 2020-02-27; First posted 2020-03-17 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Eosinophilic Esophagitis; Diagnoses Disease
Keywords: eosinophilic esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- EoE patients (Other): Patients will all be administered the EsoCheck device as a diagnostic test
  Interventions: Device: EsoCheck

INTERVENTIONS:
Device: EsoCheck — All patients with known diagnosis of EoE will be administered the EsoCheck device prior to standard of care endoscopy

SUMMARY:
Eosinophilic esophagitis (EoE) is a prevalent chronic inflammatory condition of the esophagus characterized by esophageal eosinophilia that can lead to inflammation and stricture formation. To assess remission, esophagogastroduodenoscopies (EGD) with biopsies are performed. This can lead to multiple EGDs, which are invasive and costly procedures. EsoCheck is a promising noninvasive device. It is an encapsulated balloon that can be easily swallowed and collect cells from the distal esophagus. The primary aim of this study is to determine the feasibility and safety of EsoCheck compared with standard endoscopy and biopsies in the assessment of EoE. This will be a prospective cross-sectional study of adult patients (greater than or equal to 22 years of age) at the University of Pennsylvania with a diagnosis of EoE scheduled for a clinically indicated upper endoscopy.

DETAILED DESCRIPTION:
Background Eosinophilic esophagitis (EoE) is a chronic inflammatory condition of the esophagus characterized by esophageal eosinophilia that can lead to esophageal remodeling and stricture formation. To assess remission, upper endoscopy (EGD) with biopsies is performed. This is an invasive procedure and contributes to cost burden for patients. It is important to assess non-invasive techniques to sample the cells of the esophagus.

There have been a few non-invasive testing modalities suggested, including the esophageal string test and Cytosponge. These involve swallowing a string or capsule that ultimately collects esophageal cells. The string test study showed a significant correlation with traditional biopsy pathology, however, limitations included the string remaining in overnight and potential contamination from oral flora. Katzka et al showed that the Cytosponge had an 86% specificity with limitations including gelatin allergy, local esophageal abrasions and similar potential oral contamination as the esophageal string test.

Another promising device is EsoCheck. This is an encapsulated balloon that can be easily swallowed and collect cells from the distal esophagus. It is well tolerated and, in Barrett's esophagus, detected metaplasia with 91.7% specificity. The primary aims of this study are to determine the feasibility and safety of EsoCheck compared with standard endoscopy and biopsies in the assessment of EoE. Secondary aims include specific and sensitivity of EsoCheck as well as specificity and sensitivity of brush cytology given that EsoCheck is a cytology device.

Detailed Description Study design This is a prospective pilot study at the University of Pennsylvania to evaluate feasibility and safety. Inclusion criteria include patients at least 22 years of age with known EoE diagnosed in accordance with consensus guidelines previously scheduled upper endoscopy at the University of Pennsylvania. Exclusion criteria include: known or suspected contraindication for esophageal intubation, esophageal stricture with inability to pass an endoscope, history of esophageal perforation, history of esophageal resection, esophageal diverticula, esophageal fistula, pill dysphagia, pill swallowing phobia, food impaction, esophageal varices, coagulopathy, active anticoagulation or antithrombotics, active GI bleeding and pregnancy.

Consecutive patients will be approached for consent until a total of 20 patients are enrolled. Patients will be approached during the same clinic visit if they meet inclusion criteria that arranges for the EGD or via telephone up to 2 weeks prior to scheduled EGD. Charts will be reviewed and patients will be asked medical and surgical history questions to assess if any exclusion criteria. Written consent will be obtained on the day of endoscopy. Charts will be reviewed and patients called at 1 week follow up to assess if any adverse events.

EsoCheck Description The investigational product is called EsoCheck. EsoCheck is an encapsulated, inflatable, surface-textured balloon that is pill-sized (16x9mm) attached to a thin 2.16 mm silicone catheter. The device is swallowed with water. The catheter will be held without any tension to facilitate easy delivery to the stomach. The balloon is then inflated by injecting 5 cc of air through the catheter. This will be gently withdrawn until the tension from the esophageal sphincter is felt by the endoscopist. It is then pulled slowly to sample the esophagus. The balloon is then deflated while still in the distal esophagus using a syringe and inverted back into the capsule.

EsoCheck Administration and Upper Endoscopy During the intervention period of the trial, patients will arrive early for their scheduled endoscopy. This involves swallowing the balloon device while unsedated. They will then undergo their previously scheduled endoscopy with standard biopsies taken as well as brush cytology performed as EsoCheck is a cytology device to best compare histology.

EsoCheck and Brush Cytology Sample Processing and Handling:

After retrieval of the capsule through the mouth, the balloon will be re-inflated, cut from the capsule at the junction of the balloon and the holding capsule. This will be immediately placed into a pre-labeled vial of Preservcyt transport medium. Vials will be stored on site in locked cabinets at room temperature. They will be shipped in small batches with de-identified patient study numbers and sent to the Cytology Department c/o Dr. Joseph Willis, University Hospitals Cleveland Medical Center.

Specimens will be processed according to the standard operating procedures of the Department of Pathology at the University Hospitals Cleveland Medical Center. The vial containing the balloon is vortexed for 5 minutes, after which the balloon is then discarded. After centrifugation, the vial is then loaded onto the ThinPrep processor along with required assembly elements - including a pre-labeled slide corresponding to the received specimens. The ThinPrep filter rotates within the specimen vial creating turbulence that is strong enough to separate cells, debris and mucus. In cell collection, a vacuum collects cells on the exterior of the membrane of the filter. In cell transfer, the filter is inverted and gently pressed against the ThinPrep microscope slide. Slight positive air pressure causes the cells to adhere to the microscope slide resulting in an even distribution of cells in a circular area. A ThinPrep slide is then generated and is deposited in an alcohol fixative bath. The slide is then stained with a Hematoxylin and Eosin stain and cover slipped. After the ThinPrep slides are made, attempts will be made to prepare cell blocks from the reminder of the material Cytology brush samples will be analyzed at the University Hospitals Cleveland Medical Center as well with specimens processed according to the standard operating procedures.

Histologic and cytologic assessment EsoCheck derived samples will be analyzed at the University Hospitals Cleveland Medical Center. ThinPrep slidesare given to a trained gastroenterology cytopathologist for review. As the ThinPrep technology smears collected cells onto the slide in a uniform manner using a membrane-based technology, the cytopathologist will count eosinophils in one quadrant of the ThinPrep slide. These results will then be compared with the clinical and pathological features of the study individuals. The cell blocks will also be reviewed and results correlated with the ThinPrep slide results.

Assessment of brush cytology specimens will be performed at the Department of Pathology at the University Hospitals Cleveland Medical Center to include assessing eosinophil count per high power field (hpf).

Histologic assessment of esophageal biopsies will be performed as part of standard of care at the University of Pennsylvania Department of Pathology and will include assessing eosinophil count/hpf.

Surveys: Endoscopists will be surveyed regarding perceived anxiety level and comfort level during procedure. Patients will be surveyed before and afterwards regarding confidence level, anxiety level, satisfaction, willingness to undergo it again, and preference of EsoCheck compared with EGD. This survey will be repeated at a 1 week telephone follow up.

Statistical Plan: Baseline and demographic characteristics will be summarized by standard descriptive statistics (including mean and standard deviation for continuous variables such as age and standard percentages for categorical variables such as gender). The primary endpoint will be descriptive statistics of feasibility and patient safety assessed based on the answers to surveys as listed above. Secondary endpoints include the sensitivity and specificity of Esocheck with EGD and biopsy as gold standard. Secondary endpoints also include sensitivity and specificity of brush cytology with EGD and biopsy as gold standard. All subjects entered into the study will have detailed information collected on adverse events for the overall study safety analysis

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 22 years of age
* Known EoE
* Previously scheduled upper endoscopy at the University of Pennsylvania

Exclusion Criteria:

* do not meet inclusion criteria
* do not want to participate
* known or suspected contraindication for esophageal intubation
* esophageal stricture with inability to pass an endoscope
* history of esophageal perforation
* history of esophageal resection
* esophageal diverticula
* esophageal fistula
* pill dysphagia
* pill swallowing phobia
* food impaction
* esophageal varices
* coagulopathy
* active anticoagulation or antithrombotic
* active GI bleeding
* pregnancy.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-08-23 (Actual)

PRIMARY OUTCOMES:
Safety - Incidence of Adverse Events | 12 months
  One of the primary endpoints will be incidence of adverse events.This will be determined by chart review, telephone call, and any adverse events listed by endoscopist during procedure.
Feasibility - Incidence of patient being able to complete intervention of EsoCheck | 12 months
  The incidence that patient is able to complete EsoCheck. This will be determined by a yes/no survey by the endoscopist stating whether or not the patient successfully completed the intervention.

SECONDARY OUTCOMES:
Sensitivity and Specificity of EsoCheck | 12 months
  Sensitivity and specificity of Esocheck with EGD and biopsy as gold standard.
Sensitivity and Specificity of Brush Cytology | 12 months
  Sensitivity and specificity of brush cytology with EGD and biopsy as gold standard. This is an important reference as EsoCheck is a cytology device.

CONTACTS AND LOCATIONS:
Overall Officials: Gary W Falk, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lucendo AJ, Molina-Infante J, Arias A, von Arnim U, Bredenoord AJ, Bussmann C, Amil Dias J, Bove M, Gonzalez-Cervera J, Larsson H, Miehlke S, Papadopoulou A, Rodriguez-Sanchez J, Ravelli A, Ronkainen J, Santander C, Schoepfer AM, Storr MA, Terreehorst I, Straumann A, Attwood SE. Guidelines on eosinophilic esophagitis: evidence-based statements and recommendations for diagnosis and management in children and adults. United European Gastroenterol J. 2017 Apr;5(3):335-358. doi: 10.1177/2050640616689525. Epub 2017 Jan 23. PMID 28507746
- [Background] Dellon ES, Gonsalves N, Hirano I, Furuta GT, Liacouras CA, Katzka DA; American College of Gastroenterology. ACG clinical guideline: Evidenced based approach to the diagnosis and management of esophageal eosinophilia and eosinophilic esophagitis (EoE). Am J Gastroenterol. 2013 May;108(5):679-92; quiz 693. doi: 10.1038/ajg.2013.71. Epub 2013 Apr 9. PMID 23567357
- [Background] Liacouras CA, Furuta GT, Hirano I, Atkins D, Attwood SE, Bonis PA, Burks AW, Chehade M, Collins MH, Dellon ES, Dohil R, Falk GW, Gonsalves N, Gupta SK, Katzka DA, Lucendo AJ, Markowitz JE, Noel RJ, Odze RD, Putnam PE, Richter JE, Romero Y, Ruchelli E, Sampson HA, Schoepfer A, Shaheen NJ, Sicherer SH, Spechler S, Spergel JM, Straumann A, Wershil BK, Rothenberg ME, Aceves SS. Eosinophilic esophagitis: updated consensus recommendations for children and adults. J Allergy Clin Immunol. 2011 Jul;128(1):3-20.e6; quiz 21-2. doi: 10.1016/j.jaci.2011.02.040. Epub 2011 Apr 7. PMID 21477849
- [Background] Hiremath G, Gupta SK. Promising Modalities to Identify and Monitor Eosinophilic Esophagitis. Clin Gastroenterol Hepatol. 2017 Nov;15(11):1655-1664. doi: 10.1016/j.cgh.2017.05.004. Epub 2017 May 10. PMID 28501533
- [Background] Katzka DA, Geno DM, Ravi A, Smyrk TC, Lao-Sirieix P, Miremadi A, Debiram I, O'Donovan M, Kita H, Kephart GM, Kryzer LA, Camilleri M, Alexander JA, Fitzgerald RC. Accuracy, safety, and tolerability of tissue collection by Cytosponge vs endoscopy for evaluation of eosinophilic esophagitis. Clin Gastroenterol Hepatol. 2015 Jan;13(1):77-83.e2. doi: 10.1016/j.cgh.2014.06.026. Epub 2014 Jul 3. PMID 24997328
- [Background] Katzka DA, Smyrk TC, Alexander JA, Geno DM, Beitia RA, Chang AO, Shaheen NJ, Fitzgerald RC, Dellon ES. Accuracy and Safety of the Cytosponge for Assessing Histologic Activity in Eosinophilic Esophagitis: A Two-Center Study. Am J Gastroenterol. 2017 Oct;112(10):1538-1544. doi: 10.1038/ajg.2017.244. Epub 2017 Aug 15. PMID 28809387
- [Background] Furuta GT, Kagalwalla AF, Lee JJ, Alumkal P, Maybruck BT, Fillon S, Masterson JC, Ochkur S, Protheroe C, Moore W, Pan Z, Amsden K, Robinson Z, Capocelli K, Mukkada V, Atkins D, Fleischer D, Hosford L, Kwatia MA, Schroeder S, Kelly C, Lovell M, Melin-Aldana H, Ackerman SJ. The oesophageal string test: a novel, minimally invasive method measures mucosal inflammation in eosinophilic oesophagitis. Gut. 2013 Oct;62(10):1395-405. doi: 10.1136/gutjnl-2012-303171. Epub 2012 Aug 15. PMID 22895393
- [Background] Moinova HR, LaFramboise T, Lutterbaugh JD, Chandar AK, Dumot J, Faulx A, Brock W, De la Cruz Cabrera O, Guda K, Barnholtz-Sloan JS, Iyer PG, Canto MI, Wang JS, Shaheen NJ, Thota PN, Willis JE, Chak A, Markowitz SD. Identifying DNA methylation biomarkers for non-endoscopic detection of Barrett's esophagus. Sci Transl Med. 2018 Jan 17;10(424):eaao5848. doi: 10.1126/scitranslmed.aao5848. PMID 29343623
- [Background] Reed CC, Dellon ES. Eosinophilic Esophagitis. Med Clin North Am. 2019 Jan;103(1):29-42. doi: 10.1016/j.mcna.2018.08.009. Epub 2018 Nov 1. PMID 30466674
- [Background] Alexander JA, Jung KW, Arora AS, Enders F, Katzka DA, Kephardt GM, Kita H, Kryzer LA, Romero Y, Smyrk TC, Talley NJ. Swallowed fluticasone improves histologic but not symptomatic response of adults with eosinophilic esophagitis. Clin Gastroenterol Hepatol. 2012 Jul;10(7):742-749.e1. doi: 10.1016/j.cgh.2012.03.018. Epub 2012 Apr 1. PMID 22475741
- [Background] Jensen ET, Kappelman MD, Martin CF, Dellon ES. Health-care utilization, costs, and the burden of disease related to eosinophilic esophagitis in the United States. Am J Gastroenterol. 2015 May;110(5):626-32. doi: 10.1038/ajg.2014.316. Epub 2014 Sep 30. PMID 25267327
- [Background] Kim HP, Vance RB, Shaheen NJ, Dellon ES. The prevalence and diagnostic utility of endoscopic features of eosinophilic esophagitis: a meta-analysis. Clin Gastroenterol Hepatol. 2012 Sep;10(9):988-96.e5. doi: 10.1016/j.cgh.2012.04.019. Epub 2012 May 18. PMID 22610003
- [Background] van Rhijn BD, Verheij J, Smout AJ, Bredenoord AJ. The Endoscopic Reference Score shows modest accuracy to predict histologic remission in adult patients with eosinophilic esophagitis. Neurogastroenterol Motil. 2016 Nov;28(11):1714-1722. doi: 10.1111/nmo.12872. Epub 2016 Jun 2. PMID 27254480